CLINICAL TRIAL: NCT01107990
Title: Global and Regional Myocardial Strain and Power Output In Patients With Single Ventricles Using Novel MRI Techniques
Status: Terminated | Type: Observational
Why Stopped: PI time constraints
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H64391-34645-01
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Fontan Procedure; Hypoplastic Left Heart Syndrome; Tricuspid Atresia; Double Inlet Left Ventricle
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Tricuspid Atresia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Single right ventricles
- Single left ventricles

SUMMARY:
The investigators are beginning a clinical research study here at UCSF to learn more about how hearts with single ventricles work. The investigators hypothesize that myocardial strain , as measured by cardiac MRI,in patients with single ventricles differs from normal hearts. This abnormality is associated with depressed cardiac power output and impaired exercise capacity. The study will utilize cardiac magnetic resonance imaging, exercise testing, and lung function testing to study how the single ventricle heart works so that in the future the investigators can improve how the investigators care for patients with this type of congenital heart disease.

The research protocol involves: Cardiac magnetic resonance imaging (MRI of the heart), exercise tests, and lung function tests. Some of these tests are routinely used to follow patients with single ventricles. Some of these tests are part of the research protocol. If you agree to participate in this study, these tests will be performed at UCSF. The results of the routine tests will be shared with your doctor.

Participation will require approximately 30 additional minutes to the cardiac MRI procedure to collect the research data. The exercise tests, and lung function tests time commitment will take about two hours.

ELIGIBILITY:
Inclusion Criteria:

* Anatomy: The investigators will enroll 10 patients with single right ventricles status post Fontan and 10 patients with single left ventricles status post Fontan.
* Age range: 5 patients in each group will be between the ages of 10-18 years of age and 5 patients in each group will be older than 18 years of age.

Exclusion Criteria:

* Study subjects will be excluded if there are any contraindications to MRI including permanent pacemaker, ICD, retained permanent wires, cerebral aneurysm clips, neurostimulators, insulin or infusion pumps, implanted drug infusion devices, bone growth/fusion stimulators, or cochlear implants.
* In addition, patients with implanted hardware that may lead to inadequate imaging, such as steel coils or ventricular septal defect occluder devices, will be excluded.
* Finally, patients with developmental delay or physical limitations precluding cooperation with the MRI or exercise test or patients with claustrophobia will be excluded. Patients will be asked if there is any chance that they are pregnant. If they are possibly pregnant, they will be excluded.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study subjects: Patients with univentricular hearts who have undergone a Fontan procedure will be recruited for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09-20 (Actual); Study Completion 2012-09-20 (Actual)

PRIMARY OUTCOMES:
Global and regional myocardial strain (radial, longitudinal and circumferential) as measured by cardiac MRI. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lowenthal, MD, Principal Investigator — University of California, San Francisco; Alison Meadows, MD, PhD, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San-Francisco, San Francisco, California, United States